CLINICAL TRIAL: NCT05101447
Title: Pharmacokinetically-driven Dosing of Mycophenolate Mofetil for the Treatment of Pediatric Proliferative Lupus Nephritis
Acronym: PRUNE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: funding not secured
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Hermine Brunner, MD, Director, Division of Rheumatology, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRUNE
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MMF PK (Experimental)
  Interventions: Drug: Mycophenolate Mofetil
- MMF BSA (Active Comparator)
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Mycophenolate Mofetil — At baseline, subjects will be randomized 1:1 to one of two treatment arms: the current standard of clinical care [MMFBSA: 600 mg/m2/dose; max: 3 gram/day] or pharmacokinetically-driven precision dosing [MMFPK: 12-hour target area under the exposure curve of MPA (MPA-AUC0-12) at 60 mg*h/L].

SUMMARY:
Meta-analyses in adults suggest equivalence of clinical efficacy of intravenous cyclophosphamide and mycophenolate mofetil when dosed based on patient weight or body-surface-area (MMFBSA), as is the current standard for the treatment of proliferative lupus nephritis (LN) treatments in the U.S. Pharmacokinetically-guided precision dosing of MMF (MMFPK) may offer a beneficial modification of the current standard treatment in that MMKPK promises over 30% higher LN response rates than MMFBSA. The objective of the proposed randomized, controlled study is to compare the efficacy and safety of pharmacokinetically-guided precision dosing of MMF (MMFPK) with conventional dosing regimens of MMF (MMFBSA) among children with proliferative LN.

ELIGIBILITY:
Inclusion Criteria:

New diagnosis with proliferative LN based on kidney biopsy done within 4 weeks of enrollment Diagnosis with childhood-onset SLE (cSLE) as per the ACR criteria95, 96 Age 8 - 17 years at the time of enrollment96 Tolerates oral MMF

Exclusion Criteria:

Perceived or stated inability to adhere to study protocol, Lack of use of highly effective birth control method. Presence of cSLE features that a-priori suggest that the patient benefits from other therapy than that suggested by the study protocol, History of significant kidney disease prior to the diagnosis with cSLE, Need for renal replacement therapy at the time of enrolment, Concurrent therapy with CYC or rituximab.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
renal remission | 26 week
  defined as at least PRR (CRR or PRR)

SECONDARY OUTCOMES:
Complete Renal Remission | week 26
  CRR

IPD SHARING:
Plan to Share IPD: Undecided